CLINICAL TRIAL: NCT07403344
Title: Comparative Effects of Sahrmann and Kendall Exercises on Pain, Range of Motion and Disability in Patients With Text Neck Syndrome.
Brief Title: Comparative Effects of Sahrmann and Kendall Exercises in Patients With Text Neck Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0183
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Text Neck Syndrome
Keywords: Disability; Neck pain; Range of motion; Kendall exercise; Sahrmann exercise
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sahrmann exercise (Experimental)
  Interventions: Other: Sahrmann exercise; Other: Standard Physical Therapy Treatment
- Kendall Exercise (Active Comparator)
  Interventions: Other: Kendall exercise; Other: Standard Physical Therapy Treatment

INTERVENTIONS:
Other: Sahrmann exercise — Sahrmann exercises which include Deep Neck Flexor Activation (Chin Tucks), Cervical Flexion with Scapular Stabilization, Shoulder Blade Retractions, Controlled Cervical Rotations, Scapular Depression with Resistance Bands, Neck Flexion Isometric, Cervical Side Bending with Resistance, Thoracic Extension Exercises. Each containing 5 repetitions, each held for 5-10 seconds, Total 3 sessions per week for 4 weeks.
  Arms: Sahrmann exercise
Other: Kendall exercise — Kendall exercise includes Deep Neck Flexor Activation (supine chin tucks) for 2 to 8s, stretch cervical extensors, Scapular Retraction with resistance, Pectoralis major and minor stretch. Each posture was maintained for 30s and 6 sets of 12 repetitions were performed with 3 sessions per week on alternate days for 4 weeks.
  Arms: Kendall Exercise
Other: Standard Physical Therapy Treatment — Both groups were given Standard Physical Therapy treatment including hot pack (applying a moist heat pack to the neck for 7-10 minutes, relaxing muscles, and alleviating pain. Use a towel as a barrier to avoid burns.) and Soft Tissue Mobilization Protocol (involves applying targeted pressure to neck muscles, releasing tension and improving circulation. Additionally, postural education focused on maintaining an upright posture while using mobile devices. This involved holding the device close to eye level and using it while either standing or sitting. Repeat 2-3 times daily for 4 weeks.

SUMMARY:
The study was conducted to determine the comparative effects of Sahrmann and Kendall exercises on pain, range of motion and disability in patients with text neck syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 35 years
* Both male and female were included.
* Participants who used smartphone for more than 2 hours daily
* Participant with neck pain aggravated by sustained posture, stiffness on neck and neck turning, the Craniovertebral angle (CVA) <50°
* Participant with rounded shoulder angle (RSA) greater than 52° (51)
* Participants with pain greater than 5 on numeric pain rating scale (NPRS)
* Participants with neck disability index (NDI) of >10

Exclusion Criteria:

* • Participants with any spinal infection example: osteomyelitis

  * Participant with any inflammatory condition example: rheumatoid arthritis
  * Participant with any previous cervical surgery
  * Traumatic injury
  * Torticollis, and scoliosis or any pregnant females
  * Participant with any disc prolapse or other spinal issues like stenosis, herniation of disc, spondylolisthesis and osteoporosis
  * Participants taking pain related medication or have gone under physical therapy sessions
  * Participant with Malignancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment to the end of treatment at 4 weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Neck Disability Index | From enrollment to the end of treatment at 4 weeks
  Neck pain disability index is used for the disability of the neck or the impact of neck pain on a person. This 10-item questionnaire is used to assess the patient overall quality of life as well as the personal ability to perform activities of daily living. It has various categories ranging from personal care, lifting, reading etc. it has a scoring range from zero disability. The greater the scored the higher the disability of neck.

SECONDARY OUTCOMES:
ROM Cervical Spine (Flexion) | From enrollment to the end of treatment at 4 weeks
  Changes in cervical spine flexion ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Extension) | From enrollment to the end of treatment at 4 weeks
  Changes in cervical spine extension ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Lateral Flexion) Left Side | From enrollment to the end of treatment at 4 weeks
  Changes in cervical spine Lateral flexion on left side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (lateral Flexion) Right Side | From enrollment to the end of treatment at 4 weeks
  Changes in cervical spine lateral flexion on right side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Left Side | From enrollment to the end of treatment at 4 weeks
  Changes in cervical spine rotation on left side ROM at baseline and 4th week of intervention was measured using goniometer.
ROM Cervical Spine (Rotation) Right Side | From enrollment to the end of treatment at 4 weeks
  Changes in cervical spine rotation on right side ROM at baseline and 4th week of intervention was measured using goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- PulseCore Physio and Rehab Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Letafatkar A, Rabiei P, Alamooti G, Bertozzi L, Farivar N, Afshari M. Effect of therapeutic exercise routine on pain, disability, posture, and health status in dentists with chronic neck pain: a randomized controlled trial. Int Arch Occup Environ Health. 2020 Apr;93(3):281-290. doi: 10.1007/s00420-019-01480-x. Epub 2019 Oct 25. PMID 31654125
- [Background] Jabbar KM, Gandomi F. The comparison of two corrective exercise approaches for hyperkyphosis and forward head posture: A quasi-experimental study. J Back Musculoskelet Rehabil. 2021;34(4):677-687. doi: 10.3233/BMR-200160. PMID 33896809
- [Background] Abdel-Aziem AA, Mohamed RR, Draz AH, Azab AR, Hegazy FA, Diab RH. The effect of McKenzie protocol vs. deep neck flexor and scapulothoracic exercises in subjects with chronic neck pain - a randomized controlled study. Eur Rev Med Pharmacol Sci. 2022 May;26(9):3138-3150. doi: 10.26355/eurrev_202205_28731. PMID 35587064
- [Background] Abu-Taleb W, Yamany AA, Aneis YM, Abu El Kasem ST. Effect of adding global postural reeducation to kendall exercises for treating asymptomatic forward head posture: A single-blinded randomized controlled trial. J Bodyw Mov Ther. 2025 Jun;42:938-947. doi: 10.1016/j.jbmt.2025.01.039. Epub 2025 Feb 6. PMID 40325777